CLINICAL TRIAL: NCT05761197
Title: Association Between Early Candida Infection (Oral Thrush) and Severe Early Childhood Caries (S-ECC)
Brief Title: Oropharyngeal Candidiasis (OPC) and S-ECC
Acronym: Oral-Thrush
Status: Recruiting | Type: Observational
Sponsor: Temple University (Other)
Collaborators: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Other Study IDs: 31690
Record Dates: First submitted 2023-02-22; First posted 2023-03-09 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Candida Infection; Oral Thrush; Early Childhood Caries
Keywords: Oral candidiasis; Candida infection; Oral thrush; Early childhood caries; Oral Health
MeSH Terms: conditions — Candidiasis; Candidiasis, Oral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children with history of OPC: Individuals in the non-OPC cohort will be age and sex-matched to individuals in the OPC cohort.
- Children without history of OPC: Individuals in the OPC cohort will be age and sex-matched to individuals in the non-OPC cohort.

SUMMARY:
The overall objective of this study is to investigate the association of early Candida infection (known as oral thrush or oropharyngeal candidiasis, OPC) in children during the first year of life with the onset and severity of severe early childhood caries (S-ECC).

DETAILED DESCRIPTION:
The overall goal of this study is to conduct a longitudinal observational study to investigate the association of early OPC with the onset and severity of S-ECC to better understand the role of Candida (particularly C. albicans) in severe childhood caries. The investigators will test the hypothesis that OPC is associated with S-ECC by modifying the plaque microbiota and enhancing virulence in a manner that is conducive to the early development of the disease.

For this study, a total of 70 infants (aged 9-15-month-old) with or without a history of OPC in their first year of life will be enrolled, based on the inclusion and exclusion criteria. Subjects will have their medical/dental history reviewed from medical records. At each study visit (Baseline, 6-month, 12-month, 18-month, and 24-month follow-ups), an oral examination including soft tissue and caries exam will be performed by a calibrated evaluator. Dental plaque/oral swab samples will be collected at each study visit. In addition, a comprehensive survey including demographic status, oral hygiene, diet, delivery, and feeding method as well as current medication usage will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Male or female individuals at the age of 9-24-month-old
* Must have at least one fully erupted tooth at baseline visit
* Parent/guardian willing and able to provide informed consent
* With or without a history of OPC (the study team will enroll 35 participants with and 35 participants without a history of OPC)

Exclusion Criteria:

* Presence of a systemic medical condition (e.g. Down syndrome etc.)
* Presence of an orofacial deformity
* Presence of dental caries
* Use of systemic antimicrobial therapy within 30 days of the baseline visit
* Presence of any condition which, in the opinion of the investigator, makes participation in the project not in the individual's best interest.

Ages: 9 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study team will recruit 70 subjects (35 subjects with a history of OPC and 35 subjects without a history of OPC) for this study.
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
To explore the association between OPC and S-ECC onset and severity | 24 months
  Caries will be measured by ICDAS scoring system; Plaque and oral swab samples will be collected at each study visit (Baseline, 6-month, 12-month,18-month and 24-month follow-ups); Candida strains will be detected using culturing-dependent and -independent sequencing techniques.

SECONDARY OUTCOMES:
To evaluate the influence of OPC on the oral microbiota | 24 months
  Microbiome profiling will be done by shot gun sequencing

OTHER OUTCOMES:
To study the role of Candida on biofilm cariogenic properties | 24 months
  Candida-bacterial interaction in modulating biofilm development and virulence will be evaluated using validated experimental models

CONTACTS AND LOCATIONS:
Overall Officials: Yuan Liu, DDS, MS, PhD, Principal Investigator — Temple University Kornberg School of Dentistry
Locations (1):
- Temple University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kassebaum NJ, Smith AGC, Bernabe E, Fleming TD, Reynolds AE, Vos T, Murray CJL, Marcenes W; GBD 2015 Oral Health Collaborators. Global, Regional, and National Prevalence, Incidence, and Disability-Adjusted Life Years for Oral Conditions for 195 Countries, 1990-2015: A Systematic Analysis for the Global Burden of Diseases, Injuries, and Risk Factors. J Dent Res. 2017 Apr;96(4):380-387. doi: 10.1177/0022034517693566. PMID 28792274
- [Background] GBD 2016 Disease and Injury Incidence and Prevalence Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 328 diseases and injuries for 195 countries, 1990-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet. 2017 Sep 16;390(10100):1211-1259. doi: 10.1016/S0140-6736(17)32154-2. PMID 28919117
- [Background] Hajishengallis E, Parsaei Y, Klein MI, Koo H. Advances in the microbial etiology and pathogenesis of early childhood caries. Mol Oral Microbiol. 2017 Feb;32(1):24-34. doi: 10.1111/omi.12152. Epub 2016 Feb 4. PMID 26714612
- [Background] Bowen WH, Burne RA, Wu H, Koo H. Oral Biofilms: Pathogens, Matrix, and Polymicrobial Interactions in Microenvironments. Trends Microbiol. 2018 Mar;26(3):229-242. doi: 10.1016/j.tim.2017.09.008. Epub 2017 Oct 30. PMID 29097091
- [Background] Hajishengallis E, Forrest CB, Koo H. Early Childhood Caries: Future Perspectives in Risk Assessment. JDR Clin Trans Res. 2016 Jul;1(2):110-111. doi: 10.1177/2380084416637577. Epub 2016 Mar 7. No abstract available. PMID 28879240
- [Background] American Academy on Pediatric Dentistry; American Academy of Pediatrics. Policy on early childhood caries (ECC): classifications, consequences, and preventive strategies. Pediatr Dent. 2008-2009;30(7 Suppl):40-3. No abstract available. PMID 19216381
- [Background] de Carvalho FG, Silva DS, Hebling J, Spolidorio LC, Spolidorio DM. Presence of mutans streptococci and Candida spp. in dental plaque/dentine of carious teeth and early childhood caries. Arch Oral Biol. 2006 Nov;51(11):1024-8. doi: 10.1016/j.archoralbio.2006.06.001. Epub 2006 Aug 7. PMID 16890907
- [Background] Raja M, Hannan A, Ali K. Association of oral candidal carriage with dental caries in children. Caries Res. 2010;44(3):272-6. doi: 10.1159/000314675. Epub 2010 May 27. PMID 20516688
- [Background] Yang XQ, Zhang Q, Lu LY, Yang R, Liu Y, Zou J. Genotypic distribution of Candida albicans in dental biofilm of Chinese children associated with severe early childhood caries. Arch Oral Biol. 2012 Aug;57(8):1048-53. doi: 10.1016/j.archoralbio.2012.05.012. Epub 2012 Jun 18. PMID 22717324
- [Background] Qiu R, Li W, Lin Y, Yu D, Zhao W. Genotypic diversity and cariogenicity of Candida albicans from children with early childhood caries and caries-free children. BMC Oral Health. 2015 Nov 17;15(1):144. doi: 10.1186/s12903-015-0134-3. PMID 26576955
- [Background] Xiao J, Moon Y, Li L, Rustchenko E, Wakabayashi H, Zhao X, Feng C, Gill SR, McLaren S, Malmstrom H, Ren Y, Quivey R, Koo H, Kopycka-Kedzierawski DT. Candida albicans Carriage in Children with Severe Early Childhood Caries (S-ECC) and Maternal Relatedness. PLoS One. 2016 Oct 14;11(10):e0164242. doi: 10.1371/journal.pone.0164242. eCollection 2016. PMID 27741258
- [Background] Duangthip D, D D. Early childhood caries and candida albicans. Evid Based Dent. 2018 Dec;19(4):100-101. doi: 10.1038/sj.ebd.6401337. PMID 30573860
- [Background] Xiao J, Huang X, Alkhers N, Alzamil H, Alzoubi S, Wu TT, Castillo DA, Campbell F, Davis J, Herzog K, Billings R, Kopycka-Kedzierawski DT, Hajishengallis E, Koo H. Candida albicans and Early Childhood Caries: A Systematic Review and Meta-Analysis. Caries Res. 2018;52(1-2):102-112. doi: 10.1159/000481833. Epub 2017 Dec 21. PMID 29262404
- [Background] Metwalli KH, Khan SA, Krom BP, Jabra-Rizk MA. Streptococcus mutans, Candida albicans, and the human mouth: a sticky situation. PLoS Pathog. 2013;9(10):e1003616. doi: 10.1371/journal.ppat.1003616. Epub 2013 Oct 17. No abstract available. PMID 24146611
- [Background] Koo H, Bowen WH. Candida albicans and Streptococcus mutans: a potential synergistic alliance to cause virulent tooth decay in children. Future Microbiol. 2014;9(12):1295-7. doi: 10.2217/fmb.14.92. No abstract available. PMID 25517895
- [Background] Falsetta ML, Klein MI, Colonne PM, Scott-Anne K, Gregoire S, Pai CH, Gonzalez-Begne M, Watson G, Krysan DJ, Bowen WH, Koo H. Symbiotic relationship between Streptococcus mutans and Candida albicans synergizes virulence of plaque biofilms in vivo. Infect Immun. 2014 May;82(5):1968-81. doi: 10.1128/IAI.00087-14. Epub 2014 Feb 24. PMID 24566629
- [Background] Hwang G, Liu Y, Kim D, Li Y, Krysan DJ, Koo H. Candida albicans mannans mediate Streptococcus mutans exoenzyme GtfB binding to modulate cross-kingdom biofilm development in vivo. PLoS Pathog. 2017 Jun 15;13(6):e1006407. doi: 10.1371/journal.ppat.1006407. eCollection 2017 Jun. PMID 28617874
- [Background] Kim D, Sengupta A, Niepa TH, Lee BH, Weljie A, Freitas-Blanco VS, Murata RM, Stebe KJ, Lee D, Koo H. Candida albicans stimulates Streptococcus mutans microcolony development via cross-kingdom biofilm-derived metabolites. Sci Rep. 2017 Jan 30;7:41332. doi: 10.1038/srep41332. PMID 28134351
- [Background] Koo H, Andes DR, Krysan DJ. Candida-streptococcal interactions in biofilm-associated oral diseases. PLoS Pathog. 2018 Dec 13;14(12):e1007342. doi: 10.1371/journal.ppat.1007342. eCollection 2018 Dec. No abstract available. PMID 30543717
- [Background] Kim HE, Liu Y, Dhall A, Bawazir M, Koo H, Hwang G. Synergism of Streptococcus mutans and Candida albicans Reinforces Biofilm Maturation and Acidogenicity in Saliva: An In Vitro Study. Front Cell Infect Microbiol. 2021 Feb 19;10:623980. doi: 10.3389/fcimb.2020.623980. eCollection 2020. PMID 33680985
- [Background] Jean J, Goldberg S, Khare R, Bailey LC, Forrest CB, Hajishengallis E, Koo H. Retrospective Analysis of Candida-related Conditions in Infancy and Early Childhood Caries. Pediatr Dent. 2018 Mar 15;40(2):131-135. PMID 29663914
- [Background] Kressin NR, Nunn ME, Singh H, Orner MB, Pbert L, Hayes C, Culler C, Glicken SR, Palfrey S, Geltman PL, Cadoret C, Henshaw MM. Pediatric clinicians can help reduce rates of early childhood caries: effects of a practice based intervention. Med Care. 2009 Nov;47(11):1121-8. doi: 10.1097/MLR.0b013e3181b58867. PMID 19786919
- [Background] Hedrick VE, Comber DL, Estabrooks PA, Savla J, Davy BM. The beverage intake questionnaire: determining initial validity and reliability. J Am Diet Assoc. 2010 Aug;110(8):1227-32. doi: 10.1016/j.jada.2010.05.005. PMID 20656099
- [Background] Broffitt B, Levy SM, Warren J, Cavanaugh JE. Factors associated with surface-level caries incidence in children aged 9 to 13: the Iowa Fluoride Study. J Public Health Dent. 2013 Fall;73(4):304-10. doi: 10.1111/jphd.12028. Epub 2013 Jul 26. PMID 23889610
- [Background] Gugnani N, Pandit IK, Srivastava N, Gupta M, Sharma M. International Caries Detection and Assessment System (ICDAS): A New Concept. Int J Clin Pediatr Dent. 2011 May-Aug;4(2):93-100. doi: 10.5005/jp-journals-10005-1089. Epub 2010 Apr 15. PMID 27672245
- [Background] Shoaib L, Deery C, Ricketts DN, Nugent ZJ. Validity and reproducibility of ICDAS II in primary teeth. Caries Res. 2009;43(6):442-8. doi: 10.1159/000258551. Epub 2009 Nov 12. PMID 19907175
- [Background] Policy on Early Childhood Caries (ECC): Classifications, Consequences, and Preventive Strategies. Pediatr Dent. 2016 Oct;38(6):52-54. No abstract available. PMID 27931420
- [Background] Drury TF, Horowitz AM, Ismail AI, Maertens MP, Rozier RG, Selwitz RH. Diagnosing and reporting early childhood caries for research purposes. A report of a workshop sponsored by the National Institute of Dental and Craniofacial Research, the Health Resources and Services Administration, and the Health Care Financing Administration. J Public Health Dent. 1999 Summer;59(3):192-7. doi: 10.1111/j.1752-7325.1999.tb03268.x. No abstract available. PMID 10649591
- See also: The Global Burden of Disease 2015 study aims to use all available data of sufficient quality to generate reliable and valid prevalence, incidence, and disability-adjusted life year (DALY) estimates of oral conditions for the period of 1990 to 2015. — https://pubmed.ncbi.nlm.nih.gov/28792274/
- See also: As mortality rates decline, life expectancy increases, and populations age, non-fatal outcomes of diseases and injuries are becoming a larger component of the global burden of disease. The Global Burden of Diseases, Injuries, and Risk Factors Study 2016 — https://pubmed.ncbi.nlm.nih.gov/28919117/
- See also: This review provides a broader perspective about the etiology and pathogenesis of ECC based on previous and current knowledge on biofilm matrix, microbial diversity — https://pubmed.ncbi.nlm.nih.gov/26714612/
- See also: The article discusses recent advances in the role of the biofilm matrix and interactions between opportunistic pathogens and commensals in the pathogenesis of dental caries. — https://pubmed.ncbi.nlm.nih.gov/29097091/
- See also: Early identification and early application of preventive measures are essential to help eliminate this costly and painful disease — https://pubmed.ncbi.nlm.nih.gov/28879240/
- See also: AAPD encourages healthcare providers and caregivers to implement preventive practices that can decrease a child's risks of developing this preventable disease to reduce the burden on the child, the family, and society — https://pubmed.ncbi.nlm.nih.gov/19216381/
- See also: This study determined the presence of mutans streptococci and Candida spp. in supragingival dental plaque and infected dentine of caries-free children, with early childhood caries and caries — https://pubmed.ncbi.nlm.nih.gov/16890907/
- See also: This study was carried out to identify association between oral candidal carriage in children and dental caries. — https://pubmed.ncbi.nlm.nih.gov/20516688/
- See also: In this study, the authors investigate the presence and genotypic distribution of C. albicans in the dental biofilm of Chinese children with severe early childhood caries (S-ECC). — https://pubmed.ncbi.nlm.nih.gov/22717324/
- See also: This study aimed to explore the genotypic diversity and cariogenicity of C. albicans from children with early childhood caries and caries-free children. — https://pubmed.ncbi.nlm.nih.gov/26576955/
- See also: The goal of this study was to examine the C. albicans carriage in children with severe early childhood caries (S-ECC) and the maternal relatedness. — https://pubmed.ncbi.nlm.nih.gov/27741258/
- See also: Children with oral C. albicans have higher odds of experiencing ECC, compared to children without C. albicans. — https://pubmed.ncbi.nlm.nih.gov/30573860/
- See also: This systematic review indicates that children with oral C. albicans have >5 times higher odds of having ECC compared to those without C. albicans. — https://pubmed.ncbi.nlm.nih.gov/29262404/
- See also: The presence of C. albicans in the oral environment can now be considered an additional factor that needs to be taken into account in evaluating risks to caries — https://pubmed.ncbi.nlm.nih.gov/24146611/
- See also: The authors suggest the need to explore how Candida infection is acquired and whether some strains are more infectious than others. — https://pubmed.ncbi.nlm.nih.gov/25517895/
- See also: Using a rodent model, the authors explored the implications of the cross-kingdom interaction for the pathogenesis of dental caries. — https://pubmed.ncbi.nlm.nih.gov/24566629/
- See also: Enhanced understanding of GtfB-Candida interactions may provide new perspectives for devising effective therapies to disrupt this cross-kingdom relationship associated with an important childhood oral disease. — https://pubmed.ncbi.nlm.nih.gov/28617874/
- See also: This study was conducted to investigate how microbial products from this cross-kingdom association modulate S. mutans build-up in biofilms. — https://pubmed.ncbi.nlm.nih.gov/28134351/
- See also: Clinical data, together with in vivo studies, provide compelling evidence of the importance of cross-kingdom interactions in the severity of mucosal diseases and dental caries. — https://pubmed.ncbi.nlm.nih.gov/30543717/
- See also: The authors provide feasible data to support the clinical findings in regards to the synergistic association between S. mutans and C. albicans in the pathogenesis of ECC. — https://pubmed.ncbi.nlm.nih.gov/33680985/
- See also: The purpose of this study was to assess whether there is an association between oral thrush or other Candida-related conditions in infancy and early childhood caries (ECC) diagnosed by pediatricians. — https://pubmed.ncbi.nlm.nih.gov/29663914/
- See also: Early childhood caries (ECC) is a serious and preventable disease which pediatric clinicians can help address by counseling to reduce risk. — https://pubmed.ncbi.nlm.nih.gov/19786919/
- See also: The purpose of this cross-sectional investigation was to determine the validity and reliability of a self-administered beverage intake questionnaire (BEVQ) that estimates mean daily intake of beverages consumed across 19 beverage categories. — https://pubmed.ncbi.nlm.nih.gov/20656099/
- See also: As dental caries can progress throughout a person's lifetime, understanding caries risk factors unique to specific life phases is important. This study aims to assess caries incidence and risk factors for young adolescents. — https://pubmed.ncbi.nlm.nih.gov/23889610/
- See also: The ICDAS criteria was developed by an international team of caries researchers to integrate several new criteria systems into one standard system for caries detection and assessment. — https://pubmed.ncbi.nlm.nih.gov/27672245/
- See also: The aim of this in vitro study was to assess the validity and reproducibility of the ICDAS II (International Caries Detection and Assessment System) criteria in primary teeth. — https://pubmed.ncbi.nlm.nih.gov/19907175/
- See also: The American Academy of Pediatric Dentistry (AAPD) encourages healthcare providers and caregivers to implement preventive practices that can decrease a child's risks of developing this disease. — https://pubmed.ncbi.nlm.nih.gov/27931420/
- See also: The workshop's goal was to review current methods of diagnosis of dental caries in primary teeth and to propose case definitions and diagnostic criteria for future research projects regarding dental caries in preschool-aged children. — https://pubmed.ncbi.nlm.nih.gov/10649591/

DOCUMENTS (1):
  • Informed Consent Form (2022-08-25): https://cdn.clinicaltrials.gov/large-docs/97/NCT05761197/ICF_000.pdf